CLINICAL TRIAL: NCT06750731
Title: Real World Study of Efficacy and Adherence to Subcutaneous vs. Intravenous Vedolizumab in Patients With Inflammatory Bowel Disease Using a Novel Remote MONITORing Intervention (MONITOR Study)
Brief Title: Study of Efficacy and Adherence to Subcutaneous vs. Intravenous Vedolizumab in Patients With Inflammatory Bowel Disease Using a Novel Remote MONITORing Intervention
Acronym: MONITOR
Status: Recruiting | Type: Observational
Sponsor: Mercy Medical Center (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Raymond Cross, Director Center for Inflammatory Bowel and Colorectal Diseases, Mercy Medical Center
Other Study IDs: MMC#2024-34; IISR-2024-200548 (Other Grant/Funding Number: Takeda)
Record Dates: First submitted 2024-12-02; First posted 2024-12-27 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Inflammatory Bowel Disease (IBD); Crohn's Disease; Ulcerative Colitis
Keywords: inflammatory bowel disease; ulcerative colitis; Crohn's disease; remote monitoring; vedolizumab; Entvyio; adherence
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with IBD receiving vedolizumab
  Interventions: Device: Tappt

INTERVENTIONS:
Device: Tappt — Tappt is a web-based system designed to record participants medication taking behavior and bowel symptoms. Participants will be assigned smart labels for their specific vedolizumab regimen, which will be used by participants to record their vedolizumab use. Participants will be shipped smart labels to be affixed to an IV "card" for the first three infusions and for subsequent infusions or injections. At the time of a vedolizumab dose, participants will scan the smart label by tapping it with their mobile device to verify that they are taking the medication. Each day that vedolizumab is due, patients will receive a reminder through SMS message. If participants fail to scan the label at a given time (as expected by their specific medication regimen), they will receive an end of day text message reminder. Participants will also complete a patient reported outcome assessment at baseline, weekly for 6 weeks, and then monthly for the entire 22 weeks of the study triggered by the system.

SUMMARY:
The goal of this observational study is to assess the feasibility and effectiveness of a remote monitoring digital health system on adherence, clinical outcomes, and healthcare utilization in patients with inflammatory bowel disease (Crohn's disease, ulcerative colitis, and inflammatory bowel disease type undetermined) initiating therapy with vedolizumab (Entvyio). The main questions it aims to answer are:

1. Assess and compare adherence to intravenous (IV) and subcutaneous vedolizumab maintenance therapy in patients with IBD using a novel remote monitoring system.
2. Assess symptom response to vedolizumab post induction (week 6-8) and during maintenance therapy (week 22) using a novel remote monitoring system.
3. Assess time to response to vedolizumab during induction (weeks 0-6) using a novel remote monitoring system.

Researchers will compare medication adherence between participants using IV and subcutaneous vedolizumab maintenance therapy to see if adherence is lower with self-administration.

Participants will be asked to register adherence to medication using the novel remote monitoring system each time they take a dose of vedolizumab and to respond to two questions about bowel symptoms weekly for the first 6 weeks after starting vedolizumab then monthly thereafter for 6 months. Additionally, participants will be asked to enter information regarding demographics and social determinants of health at baseline and other variables listed below at baseline and at weeks 2, 6, 14, and 22 post baseline unless otherwise denoted:

* MARS-5
* Healthcare utilization (22 weeks only)
* Harvey Bradshaw Index (Crohn's disease only)
* Simple clinical colitis activity index (Ulcerative colitis only)
* PROMIS Global Health Scale
* PROMIS Anxiety
* PROMIS Depression
* PROMIS Sleep Disturbance
* PROMIS Pain Interference
* PROMIS Physical Function
* IBD Self-Efficacy
* Attitudinal Survey (22 weeks only)

DETAILED DESCRIPTION:
The proposed study is a multicenter, open label, clinical trial to be conducted over 22 weeks. Participants will verify medication adherence using the Tappt web-based system. Additionally, participants will complete a two-item assessment of symptoms at baseline, weekly for 6 weeks, then monthly through week 22.

All participants are required to complete electronic data entry forms at baseline, 2, 6, 14, and 22 weeks. Adherence, disease activity, quality of life, PROs, and IBD self-efficacy will be measured at each time point during the 22-week study. Health care utilization will be measured at 22 weeks. Demographic and clinical information will be collected at the baseline visit. Questions regarding social determinants of health will be assessed at baseline.

Participants will be recruited for this study from seven clinical centers: Capital Digestive Care, MMC (lead site), New York University, Tulane University, University of North Carolina (data management center), University of Cincinnati, and Vanderbilt University. Of note, New York University has access to a disadvantaged population at NYC Health + Hospitals / Bellevue and a community site on Long Island.

Patients with an ostomy will be excluded since calculation of bowel movement frequency is not possible in this setting. For similar reasons, investigators will exclude patients who have undergone total or subtotal colectomy and/or that have short bowel syndrome. In these patients, clinical symptoms are less reliable to distinguish quiescent from active disease. Active disease will not be required for entry into the study.

All the participant's concomitant medications will be continued during the study. Addition of new IBD medications will be allowed during the study. If the new medication replaces vedolizumab, the replacement medication will be similarly tracked.

Investigators will attempt to minimize measurement bias by collecting outcomes data through electronic data capture directly from participants.

Eligible patients will complete informed consent and a baseline survey gathering demographic and clinical information. The research team will input the participant's information into the Tappt web-based system. The research team will then assign smart labels to the participant's vedolizumab regimen, which will be used by participants to record their vedolizumab use. Participants will be shipped smart labels to be affixed to an IV "card" for the first three infusions and for subsequent every 8 week infusions or every 2 week subcutaneous pen. The participant will receive sufficient labels for dosing of 154 days (22 weeks), plus additional labels to account for lost or damaged labels and dose escalation. Changes in dose of vedolizumab will be monitored on a biweekly basis by study coordinators. Any change in dosing will be updated on the Tappt web-based system; additional labels will not be required as participants are given enough labels to account for dose escalation during the study period. Participants will receive written materials and virtual training on how to attach and use the proprietary labels, set up their profile, use the patient-facing web app, and seek technical helpdesk support.

At the time of a vedolizumab dose, participants will scan the smart label by tapping it with their mobile device to verify that they are taking the medication. Upon scanning, participants immediately will receive a notification on their device indicating that the label was successfully scanned, and that their medication adherence was updated in their profile. Each day that vedolizumab is due, participants will receive a reminder through SMS message. If participants fail to scan the label at a given time (as expected by their specific medication regimen), participants will receive an end of day text message reminder. Participants will also have a "grace period" to record the doses within 3 days of the scheduled subcut regimen, and 7 days within their IV regimen, and would still be considered adherent to their schedule. If the participant did not record a dose at the completion of their grace period, they will receive a text message prompting them to respond to a survey on the reason they missed their dose. Participants will also complete a patient reported outcome (PRO) 2 assessment at baseline, weekly for 6 weeks, and then monthly for the entire 22 weeks of the study triggered by the Tappt platform, through an HTML link sent to participants by SMS message. The research team will also be able to send the PRO2 survey to participants at any given time, at their discretion, if participants are experiencing a flare or at the time of a change in vedolizumab dose or change in advanced therapy. Items for the PRO 2 vary based on disease type. The web app offers participants visibility into their medication adherence patterns and upcoming doses, as well as the opportunity to respond to questions related to PROs or reasons they have missed their doses. The system's algorithms send participants personalized alerts and reminders to help them stay engaged in care.

Two missed doses of subcut vedolizumab within 28 days and one missed dose of IV vedolizumab within 8 weeks will trigger an alert. If alerts are triggered for non-adherence, a clinical nurse, pharmacist, or social worker will contact the participant to identify barriers to adherence; remediation will be initiated if possible. For participants with CD, a PRO 2 abdominal pain score of 2 (moderate) or higher and/or a liquid stool frequency of >4 will trigger an alert. For participants with UC, a rectal bleeding score of 2 and/or a stool frequency score of 2 will trigger an alert (obvious blood most of the time or blood alone pass and stool frequency >2 stools more than normal respectively). When sites receive alerts notifying them of nonadherence and/or moderate to severe bowel symptoms, they will communicate these results to the appropriate care team as well as the provider for the participant and the site principal investigator within one business day. If the participant has listed a reason(s) for nonadherence, this should be communicated as well. Once the clinical care team and provider have determined a course of action, the alert should be resolved with a response recorded in the Tappt admin portal as to the specific action taken.

Clinical teams can review their participants' data in real-time through a HIPAA-compliant provider-facing interface. To reduce monitoring burden among clinical teams, the smart algorithms also prompt automated email alerts to the clinical team when participants' adherence or PROs fall below predetermined thresholds or when a participant reports an error on their profile. These alerts can support clinical teams in following-up with patients in a timely manner to reduce risk for poor outcomes.

Tappt will also link participants to medication-specific educational material on the Crohn's and Colitis Foundation web site and educational videos for each medication class including vedolizumab as well as other topics such as wellness, nutrition, and alternative medicine.

The outcome measures below will be assessed at baseline, 6, 14, and 22 weeks after initiating treatment. All outcome measures will be captured electronically and will not require a study or office visit.

Adherence to Treatment: The primary outcome of the proposed study will be the difference in mean MPR between intravenous and subcutaneous vedolizumab during the 22-week study. The mean MPR will be calculated as follows: MPR = number days' supply of medication obtained over observation period/total number days in observation period. If a participant discontinues vedolizumab but initiates treatment with another eligible medication, the MPR will continue to be calculated. Any delay in initiating new treatment will be adjusted for in the total number of days in the observation period (i.e., if drug A is discontinued and drug B is started 2 weeks later, the total observation period will be 365-14 days or 351 days). Research coordinators will confirm data on vedolizumab use. Self-reported adherence will be assessed with the MARS-5 questionnaire. MARS-5 is a reliable and validated instrument which includes five questions; responses are ranked on a five-point scale, where 5 = never, 4 = rarely, 3 = sometimes, 2 = often and 1 = always. Scores for each item are summed to give a total score, with higher scores indicating higher levels of reported adherence.

Assessment of Disease Activity: Secondary outcomes will include response to and time to response to intravenous induction therapy with vedolizumab and response to both intravenous and subcutaneous maintenance dosing through 22 weeks. To measure disease activity in participants with CD, we will assess the Harvey Bradshaw index (HBI) without including the item on the presence of an abdominal mass. HBI scores of less than 5, 5-7, 8-16 and >16 correlate with symptomatic remission, mildly active, moderately active, and severely active symptoms, respectively. A decrease in HBI score of 3 or 4 correlates well with a symptomatic response. In addition to calculating clinical remission and response using the above measures, investigators will create an outcome of steroid-free remission/response based on whether the participant was on concurrent steroids at the time of assessment. In participants with UC and indeterminate colitis, disease activity will be assessed with the Simple Clinical Colitis Activity Index (SCCAI). A SCCAI score of <3 has been shown to correlate with symptomatic remission whereas a decrease of 2 points has been shown to correlate with a symptomatic response. Investigators will calculate steroid-free remission as above. To assess disease activity using the Tappt system, investigators will utilize the 2-item PRO 2 for CD and UC respectively. For CD, the PRO 2 score is comprised of questions regarding frequency of bowel movements in the prior week and the degree of abdominal pain. A PRO-2 score of 8, 14, and 34 correlated with a Crohn's disease activity index (CDAI) score of 150, 220, and 450 respectively. CDAI scores less than 150 are consistent with clinical remission whereas scores >220 are consistent with moderate to severe disease. In lieu of calculating a total score, an average liquid stool frequency per day of > 4 and/or an average abdominal pain score of 2 (moderate) or higher will trigger an alert. For UC and indeterminate colitis, a PRO-2 score specific for UC will be used. It is comprised of questions related to stool frequency and rectal bleeding. A score of 2 or higher for stool frequency or rectal bleeding will trigger an alert.

In addition, if available, results of quantitative c reactive protein (CRP) and fecal calprotectin (FCP) will be extracted from the medical record at each time point to assess biologic response to vedolizumab. Research staff will use the value closest to the time of assessment. CRP correlates reasonably well with endoscopic disease activity (r=0.56) and values <5 mg/dl have a negative predictive value for endoscopic disease activity of 29-61%. Likewise, FCP correlates well with endoscopic disease activity (r=0.53) but has a better negative predictive value for endoscopic disease activity using a value of <250 mcg/g (71-97%). Likewise, investigators will collect information on endoscopic activity if available. For UC and IBD type undetermined, investigators will use the Mayo Endoscopic Score (MES). The MES was modified to remove friability in the mild disease category. A MES score of 0-1 is consistent with endoscopic improvement. For participants with CD, investigators will assess endoscopic activity with the Simple Endoscopic Score (SES-CD). A score of < 3 is consistent with inactive disease, 3-6 mildly active, 7-15 moderately active, and ≥16 severely active.

investigators will also record new steroid use (oral or topical treatment) in the interval between assessments.

Healthcare Utilization: A tertiary outcome of the proposed study will be the difference in healthcare utilization between the intravenous and subcutaneous maintenance dosing regimens during the 22-week study. For healthcare utilization, investigators will use a composite endpoint including counts of hospitalizations, urgent care/emergency room visits, IBD-related surgeries, telephone calls (primary care and IBD provider), endoscopic procedures, imaging exams, and blood and stool testing. investigators will also assess new prescriptions for corticosteroids (prednisone and budesonide) at each time point. The total events will be adjusted per 100 participant years of follow up, as the two groups will be unequal in number. In addition, investigators will evaluate each outcome individually. The relatedness of hospitalization and urgent/emergency room visits to IBD care will be determined as well. Information will be obtained from participant self-report at each assessment. This approach has been validated in patients with IBD using a modification of the Canadian Community Health Survey.

Assessment of Quality of Life and Patient Reported Outcome Measures (PRO): Additional tertiary outcomes measures will include quality of life and PRO's. PROMIS is a National Institutes of Health-funded instrument that assesses the patient's self-reported health over a 7-day time period. Participants report global health, different components of physical, mental, and social health, including physical function, anxiety, depression, fatigue, sleep disturbance, and pain interference, and higher scores indicate poorer health. PROMIS scores can be group grouped as within normal limits (<55), mild (55 to <60), moderate (60 to <70), and severe (≥70) based on domain scores measured in the US general population (Kappelman, 2014; https://www.healthmeasures.net). Minimally important differences of 2 to 6 points have been reported for other disease states, including chronic pain, stroke, osteoarthritis, and cancer.49

Self-Efficacy: Self-efficacy is a perception of a patient's ability to engage in the skills necessary to master a new challenge during obstacles. An IBD-specific self-efficacy scale has been developed. The 29-item questionnaire includes questions on managing medical care, stress and emotions, symptoms and disease, and maintaining remission. Responses range from 1-Not sure at all to 10-Totally sure. Scores range from 29 to 290 with higher scores correlating with greater self-efficacy.

Social Determinants of Health: Investigators plan to include a significant proportion of participants from disadvantaged backgrounds to increase the diversity of the study population. Also, investigators plan to assess if social determinants of health impact adherence and clinical response to medical therapy overall or differentially based on delivery of maintenance treatment. Investigators will include questions on financial resource strain, food insecurity, utility needs, housing stability, transportation, and interpersonal safety questions. These components were selected in consultation with Dr. Sara Horst as her institution is implementing these questions broadly for clinical care.

Attitudinal Survey: Participants will complete a 19-item survey upon completion of the study to gather information regarding their perceptions of the Tappt system. Each item is scored from 1 to 5 (i.e., How difficult was it to use the Tappt labels to record participant's medication taking, from 1 (very difficult) to 5 (not difficult at all)?).

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age or older
2. Have documented IBD based on usual diagnostic criteria including clinical symptoms and findings from endoscopy, radiology studies, and histology
3. Initiating treatment with vedolizumab
4. Have access to a mobile smartphone (iPhone 7 or later; Android release date 2012 or later) with reliable data and/or Wi-Fi access
5. Ability to understand the protocol and provide informed consent in English or Spanish

Exclusion Criteria:

1. Inability to speak and read English or Spanish
2. Unable to comply with the study protocol including inability to access the internet and/or inadequate access to a smart device
3. Unable to access vedolizumab due to insurance restrictions
4. Unable to follow up at respective sites due to insurance restrictions or other barriers (i.e., distance from patient's home to study site)
5. Presence of an ileostomy, colostomy, ileoanal pouch anastomosis, or ileorectal anastomosis
6. Imminent surgery (within the next 60 days)
7. History of short bowel syndrome
8. Uncontrolled medical or psychiatric disease at the opinion of the investigator

   1. Degenerative neurologic condition
   2. Unstable angina
   3. Symptomatic peripheral vascular disease
   4. Malignancy within the last 2 years (excluding squamous or basal cell cancers of the skin)
   5. Poorly controlled depression, mania, and schizophrenia
   6. Serious active infection requiring antimicrobial therapy (excluding CD patients with perianal CD on antibiotics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited for this study from seven clinical centers: Capital Digestive Care, MMC (lead site), New York University, Tulane University, University of North Carolina (data management center), University of Cincinnati, and Vanderbilt University. Of note, New York University has access to a disadvantaged population at NYC Health + Hospitals / Bellevue and a community site on Long Island.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence | From enrollment to the end of the study (22 weeks).
  The primary outcome of the proposed study will be the difference in mean medication possession ratio (MPR) between intravenous and subcutaneous vedolizumab during the 22-week study. The mean MPR will be calculated as follows: MPR = number days' supply of medication obtained over observation period/total number days in observation period.
Self Reported Medication Adherence | From enrollment to the end of the study (22 weeks).
  Self-reported adherence will be assessed with the MARS-5 questionnaire. MARS-5 is a reliable and validated instrument which includes five questions; responses are ranked on a five-point scale, where 5 = never, 4 = rarely, 3 = sometimes, 2 = often and 1 = always. Scores for each item are summed to give a total score, with higher scores indicating higher levels of reported adherence.

SECONDARY OUTCOMES:
Disease Activity Crohn's Disease | From enrollment to the end of the study (22 weeks).
  Harvey Bradshaw Index (Crohn's disease only)
Healthcare Utilization | From enrollment to the end of the study (22 weeks).
  For healthcare utilization, the investigators will use a composite endpoint including counts of hospitalizations, urgent care/emergency room visits, IBD-related surgeries, telephone calls (primary care and IBD provider), endoscopic procedures, imaging exams, and blood and stool testing. We will also assess new prescriptions for corticosteroids (prednisone and budesonide). Please note that this is a composite endpoint which will include counts of all events; thus, it is a single endpoint.
Quality of Life | From enrollment to the end of the study (22 weeks).
  PROMIS Global Health Scale
  PROMIS is a National Institutes of Health-funded instrument that assesses the patient's self-reported health over a 7-day time period. Patients report global health, different components of physical, mental, and social health, including physical function, anxiety, depression, fatigue, sleep disturbance, and pain interference, and higher scores indicate poorer health. PROMIS scores can be group grouped as within normal limits (<55), mild (55 to <60), moderate (60 to <70), and severe (≥70) based on domain scores measured in the US general population (Kappelman, 2014; https://www.healthmeasures.net). Minimally important differences of 2 to 6 points have been reported for other disease states, including chronic pain, stroke, osteoarthritis, and cancer.
Anxiety | From enrollment to the end of the study (22 weeks).
  PROMIS Anxiety
  PROMIS is a National Institutes of Health-funded instrument that assesses the patient's self-reported health over a 7-day time period.48 Patients report global health, different components of physical, mental, and social health, including physical function, anxiety, depression, fatigue, sleep disturbance, and pain interference, and higher scores indicate poorer health. PROMIS scores can be grouped as within normal limits (<55), mild (55 to <60), moderate (60 to <70), and severe (≥70) based on domain scores measured in the US general population (Kappelman, 2014; https://www.healthmeasures.net). Minimally important differences of 2 to 6 points have been reported for other disease states, including chronic pain, stroke, osteoarthritis, and cancer.
Depression | From enrollment to the end of the study (22 weeks).
  PROMIS Depression
  PROMIS is a National Institutes of Health-funded instrument that assesses the patient's self-reported health over a 7-day time period.48 Patients report global health, different components of physical, mental, and social health, including physical function, anxiety, depression, fatigue, sleep disturbance, and pain interference, and higher scores indicate poorer health. PROMIS scores can be grouped as within normal limits (<55), mild (55 to <60), moderate (60 to <70), and severe (≥70) based on domain scores measured in the US general population (Kappelman, 2014; https://www.healthmeasures.net). Minimally important differences of 2 to 6 points have been reported for other disease states, including chronic pain, stroke, osteoarthritis, and cancer.
Sleep Disturbance | From enrollment to the end of the study (22 weeks).
  PROMIS Sleep Disturbance
  PROMIS is a National Institutes of Health-funded instrument that assesses the patient's self-reported health over a 7-day time period.48 Patients report global health, different components of physical, mental, and social health, including physical function, anxiety, depression, fatigue, sleep disturbance, and pain interference, and higher scores indicate poorer health. PROMIS scores can be grouped as within normal limits (<55), mild (55 to <60), moderate (60 to <70), and severe (≥70) based on domain scores measured in the US general population (Kappelman, 2014; https://www.healthmeasures.net). Minimally important differences of 2 to 6 points have been reported for other disease states, including chronic pain, stroke, osteoarthritis, and cancer.
Fatigue | From enrollment to the end of the study (22 weeks).
  PROMIS Fatigue
  PROMIS is a National Institutes of Health-funded instrument that assesses the patient's self-reported health over a 7-day time period.48 Patients report global health, different components of physical, mental, and social health, including physical function, anxiety, depression, fatigue, sleep disturbance, and pain interference, and higher scores indicate poorer health. PROMIS scores can be grouped as within normal limits (<55), mild (55 to <60), moderate (60 to <70), and severe (≥70) based on domain scores measured in the US general population (Kappelman, 2014; https://www.healthmeasures.net). Minimally important differences of 2 to 6 points have been reported for other disease states, including chronic pain, stroke, osteoarthritis, and cancer.
Pain Interference | From enrollment to the end of the study (22 weeks).
  PROMIS Pain Interference
  PROMIS is a National Institutes of Health-funded instrument that assesses the patient's self-reported health over a 7-day time period.48 Patients report global health, different components of physical, mental, and social health, including physical function, anxiety, depression, fatigue, sleep disturbance, and pain interference, and higher scores indicate poorer health. PROMIS scores can be grouped as within normal limits (<55), mild (55 to <60), moderate (60 to <70), and severe (≥70) based on domain scores measured in the US general population (Kappelman, 2014; https://www.healthmeasures.net). Minimally important differences of 2 to 6 points have been reported for other disease states, including chronic pain, stroke, osteoarthritis, and cancer.
Frailty | From enrollment to the end of the study (22 weeks).
  PROMIS Physical Function
  PROMIS is a National Institutes of Health-funded instrument that assesses the patient's self-reported health over a 7-day time period.48 Patients report global health, different components of physical, mental, and social health, including physical function, anxiety, depression, fatigue, sleep disturbance, and pain interference, and higher scores indicate poorer health. PROMIS scores can be group grouped as within normal limits (<55), mild (55 to <60), moderate (60 to <70), and severe (≥70) based on domain scores measured in the US general population (Kappelman, 2014; https://www.healthmeasures.net). Minimally important differences of 2 to 6 points have been reported for other disease states, including chronic pain, stroke, osteoarthritis, and cancer.
Self-Efficacy | From enrollment to the end of the study (22 weeks).
  IBD Self-Efficacy
  Self-efficacy is a perception of a patient's ability to engage in the skills necessary to master a new challenge during obstacles. An IBD-specific self-efficacy scale has been developed. The 29-item questionnaire includes questions on managing medical care, stress and emotions, symptoms and disease, and maintaining remission. Responses range from 1-Not sure at all to 10-Totally sure. Scores range from 29 to 290 with higher scores correlating with greater self-efficacy.
Disease activity (UC) | From enrollment to the end of the study (22 weeks).
  Simple Clinical Colitis Activity Index (Ulcerative Colitis only)
Short Disease Activity Crohn's Disease | From enrollment to the end of the study (22 weeks).
  PRO-2 for Crohn's disease
Short Disease Activity UC | From enrollment to the end of the study (22 weeks).
  PRO-2 for Ulcerative colitis
Serum Biomarker Disease Activity | From enrollment to the end of the study (22 weeks).
  C reactive protein
Fecal Biomarker Disease Activity | From enrollment to the end of the study (22 weeks).
  Fecal calprotectin
Endoscopic Disease Activity CD | From enrollment to the end of the study (22 weeks).
  Simple endoscopic score (Crohn's disease only)
Endoscopic Disease Activity UC | From enrollment to the end of the study (22 weeks).
  Mayo endoscopic score (Ulcerative Colitis only)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond K Cross, MD, MS, Principal Investigator — Mercy Medical Center
Locations (6):
- United States (6):
  - Tulane University, New Orleans, Louisiana
  - Capital Digestive Care, Chevy Chase, Maryland
  - New York University, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
The raw data will be made available to other investigators upon receipt of a written request. Release of datasets to secondary users will be subject to approval by the investigators and Takeda. All approved users will be expected to enter into a standard data use agreement. The request must include a reason for review of the data and type of dataset they wish to receive (Microsoft® Excel Spreadsheet or SAS® dataset), and a copy of an up-to-date curriculum vitae. The dataset provided will be deidentified to prevent breach of research participant confidentiality. Further, even though the dataset will be deidentified to the greatest extent possible, investigators requesting to review our data must sign an agreement that they will not attempt to obtain protected health information on research participants. In addition to the raw data, investigators will receive a list of variable and coding definitions. Other information will be provided upon request.
Time Frame: After publication of the manuscript.
Access Criteria: See plan description above.